CLINICAL TRIAL: NCT05659199
Title: Study on the Intervention of Extracorporeal Shockwave Therapy and Myofascial Release Therapy in Chronic Pelvic Pain Syndrome
Brief Title: Extracorporeal Shockwave and Myofascial Release Therapy in Chronic Pelvic Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zongda Hospital affiliated to Southeast University (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZongdaH
Record Dates: First submitted 2022-12-09; First posted 2022-12-21 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: chronic pelvic pain syndrome; extracorporeal shockwave; myofascial release therapy; surface electromyography; sympathetic skin response
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: fascia trigger point release group extracorporeal shock wave group extracorporeal shock wave and fascial trigger point release treatment group
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- extracorporeal shockwave therapy (Experimental): extracorporeal shockwave group: Patients will be treated with extracorporeal shockwave therapy (ESWT) with bladder lithotomy position, twice a week for 4 weeks, 3,000 individually with a maximum total energy flow density of 0.25 mJ/mm2, rate 3Hz each time. Extracorporeal shockwave (RUIDI.SWT001, Shenzhen, China) can provide a kind of physical spark wave energy, that will be delivered by the probe. The water sac probe will be moved slowly over the groin, perineum and crura of the penis.
  Interventions: Device: extracorporeal shockwave
- myofascial release therapy (Experimental): myofascial release group: Based on the palpation findings, pressure was applied at 1 kg/cm2 (within the patient's tolerable range depending on the individual) to the points where patients had a VAS pain score of 4 or more during palpation. Intermittent pressure will be applied for 180-210s at the tenderness until the muscle relaxed.
  Interventions: Behavioral: myofascial release
- extracorporeal shockwave combined with myofascial release therapy (Experimental): Combined therapy group: On top of the routine palpation, the combined intervention group will be then treated with extracorporeal shockwave and myofascial release therapy in identical format as that in the intervention A and B
  Interventions: Device: extracorporeal shockwave; Behavioral: myofascial release

INTERVENTIONS:
Device: extracorporeal shockwave — Patients will be treated with extracorporeal shockwave therapy (ESWT) with bladder lithotomy position, twice a week for 4 weeks, 3,000 individually with a maximum total energy flow density of 0.25 mJ/mm2, rate 3Hz each time. Extracorporeal shockwave (RUIDI.SWT001, Shenzhen, China) can provide a kind of physical spark wave energy, that will be delivered by the probe. The water sac probe will be moved slowly over the groin, perineum and crura of the penis.
  Arms: extracorporeal shockwave combined with myofascial release therapy; extracorporeal shockwave therapy
Behavioral: myofascial release — pressure was applied at 1 kg/cm2 (within the patient's tolerable range depending on the individual) to the points where patients had a VAS pain score of 4 or more during palpation. Intermittent pressure will be applied for 180-210s at the tenderness until the muscle relaxed.
  Arms: extracorporeal shockwave combined with myofascial release therapy; myofascial release therapy

SUMMARY:
The primary aims of this research are three folds: (1) To identify more relatively effective interventions for improving pain symptoms in CP/CPPS patients. (2) To ascertain the correlation between PFM elastic modulus and tenderness symptoms. This may find a more objective method of assessing efficacy. (3) To determine the correlation between the intensity of the sympathetic response and the patient's symptoms and to explore other possible pathogenetic mechanisms.

DETAILED DESCRIPTION:
Chronic prostatitis/chronic pelvic pain syndrome is a high prevalent syndrome. Previous studies showed that extracorporeal shockwave therapy and myofascial release therapy could improve quality of life in patients with Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). Theoretically, a combined therapy with extracorporeal shockwave therapy and myofascial release therapy is likely to have significant advantages in treating CP/CPPS.

ELIGIBILITY:
Inclusion Criteria:

* ① According to the National Institutes of Health classification of prostatitis[27], all male patients meet the diagnostic criteria for chronic prostatitis type IIIB/chronic pelvic pain syndrome (pain in the bladder, groin, perineal area, genitalia or lower abdomen with no significant abnormalities on urological examination);

  * Patients are aged 20-40 years;

    * Patients with Chronic pelvic pain lasting over 6 months； ④ Patients sign the informed consent form.

Exclusion Criteria:

* ① Patients with significant coagulation disorders, perineal anatomical abnormalities, hormonal abnormalities and neurological abnormalities;

  * Patients with a clear cause of pelvic pain, such as a history of previous surgery, chronic infection, trauma, prostatitis and epididymitis;

    * Patients receiving other treatments during the study; ④ Patients with any urethral pathology;

      * Patients who have had closed lumbar injections and previous lumbar surgery within six months;

        * Patients with other conditions causing pelvic pain; ⑦ Patients with contraindications to physiotherapy; ⑧ BMI>22.9

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — There is no need to confirm the self-representation of gender identity
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle surface electromyography changes | Assessments will be conducted before the intervention (T0), before the 5th intervention (T1), immediately after the 8th intervention (T2), and at the 4th week after the end of the 8th intervention (T3),assessing changes between these time points.
  Pelvic floor muscle sEMG values will be collected using the Glazer pelvic floor muscle sEMG assessment (VISHEE SA9800) Pre-resting sEMG; Tense contraction phase sEMG; Endurance contraction phase sEMG; Post-resting EMG.
National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) changes | Assessments will be conducted before the intervention (T0), before the 5th intervention (T1), immediately after the 8th intervention (T2), and at the 4th week after the end of the 8th intervention (T3),assessing changes between these time points
  Questionnaire with 13 entries, including 4 aspects: pain and discomfort symptom score, urinary symptom score, symptom impact score, quality of life score, with a total score of 0 to 43. The severity of CP/CPPS can be graded according to the total scores: mild (1-14), moderate (15-29), or severe (30-43).
  The efficacy evaluation criteria are developed with reference to the National Institutes of Health-Chronic Prostatitis Symptom Index score. Clinical control is defined as ≥ 90% decrease in the NIH-CPSI score; obvious improvement as ≥ 60% and < 89% decrease; improvement as ≥ 30% and < 59% decrease, and ineffective as < 30% decrease.

SECONDARY OUTCOMES:
Three-dimensional quantification and Shear Wave Elastography (SWE) changes | Assessments will be conducted before the intervention (T0) and at the 4th week after the end of the 8th intervention (T3),assessing change between two time points
  Trans-rectal three-dimensional ultrasound (VOLUSON E8) will be used to assess the morphological parameters of the lacunae of the levator hiatus in CP/CPPS patients, the area of the levator hiatus is situated at a depth of 2-4 cm from the perineum, where is well within the effective range of 7-4-MHz transducers.
sympathetic skin response (SSR) changes | Assessments will be conducted before the intervention (T0) and at the 4th week after the end of the 8th intervention (T3),assessing change between two time points
  SSR is a recently established method of non-invasive somatic neurography offers the advantages of both non-invasiveness and specificity, using the SA7550 FlexComp Infiniti System (Thought Technology, Canada).
  Sympathetic skin responses will be recorded with the active electrodes placed in the left palm and the reference electrodes on the dorsum of the left hand, while the patient will be in the sitting position. A channel recording from hand will be obtained simultaneously by stimulating the contralateral median nerve at the level of the wrist with a stimulation intensity at 20 mA for 0.2 ms[29]. A total of three potentials will be recorded and the mean values will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ma, Doctor, Study Director — Zhongda Hospital
Locations (1):
- Zhongda Hospital affiliated to Southeast University, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes
No datasets were generated or analyzed during the current study. The results will be published in a peer-reviewed journal upon study completion. Datasets generated or analyzed in this study will be provided by the corresponding authors upon reasonable request.
Supporting Information: Study Protocol
Time Frame: The results will be published in a peer-reviewed journal upon study completion. Datasets generated or analyzed in this study will be provided by the corresponding authors upon reasonable request.
Access Criteria: All relevant data from this study will be made available upon study completion.

REFERENCES:
- [Derived] Huang N, Qin Z, Sun W, Bao K, Zha J, Zhang P, Feng P, Zhao X, Liu M, Shi J, Ma M. Comparing the effectiveness of extracorporeal shockwave therapy and myofascial release therapy in chronic pelvic pain syndrome: study protocol for a randomized controlled trial. Trials. 2023 Oct 18;24(1):675. doi: 10.1186/s13063-023-07633-1. PMID 37853420